CLINICAL TRIAL: NCT04224298
Title: Application of White Eye Imaging Health Care System on Diagnosis of Malignant Tumors
Brief Title: Preliminary Study on Eye Features of Patients With Malignant Tumors
Status: Completed | Type: Observational
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Dr. Xue Dong, Director, Peking University Cancer Hospital & Institute
Other Study IDs: WEIS
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Feature Elongation; Cancer Patients
Keywords: Eye; Manifestations; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Based on the theory of traditional Chinese Medicine, this study collects eye features of white eyes through the White Eye Imaging Health Care System under visible light and establishes a database of eye-eye features corresponding to the disease. The computer image analysis and artificial intelligence technology are used to visualize the eye. The features were extracted and classified, and the corresponding changes in the characteristics of the traditional Chinese medicine and the disease were analyzed statistically to establish an analytical model corresponding to the disease.

DETAILED DESCRIPTION:
1. Collecting the white-eyed eye features of 500 patients with malignant tumors and 500 non-tumor patients by the white-eye shadowless imaging acquisition system under visible light, and establishing eye-catching images of malignant tumor patients and healthy people of different diseases. Feature database.
2. Based on the collected four-dimensional eye-eye diagram, using computer image analysis and artificial intelligence technology to extract and classify the eye-eye features of the white eye, and statistically analyze the correlation between the eye-eye features and the malignant tumor. The relationship between the characteristics of the white eye and the corresponding change of malignant tumor.

ELIGIBILITY:
Inclusion Criteria:

* Malignant tumor patients with clear pathological diagnosis;

  * Those who have no serious primary diseases of the cardiovascular, cerebrovascular, respiratory, endocrine, urinary, blood and other systems;

    * The main organs (hematopoiesis, heart, lung, liver, and kidney) have no obvious abnormal function; ④Age ≥18 years old, ≤75 years old; ⑤ No serious eye disease;

      * The patient volunteered to participate in this study.

Exclusion Criteria:

* Patients with severe blood loss (because when the bleeding exceeds 300ml, the white eye color of the patient is often pale white);

  * Poor patient compliance; ③ pregnant and lactating women;

    * Can't cooperate with inspection properly; ⑤ Cannot read or understand the scale.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants in the study were patients with malignant tumors and healthy volunteers.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Model of white-eye ocular features in patients with malignant tumors | 2.5 years
  The test will use Artificial Intelligence technology to analyze and learn the features of white-eye eyes of healthy people and patients with malignant tumors, and establish a model of eye characteristics of malignant tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Dong D Xue, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Yichen Dr. Xu, Beijing, China

IPD SHARING:
Plan to Share IPD: No
This research is still in the exploratory stage and there are no plans to share IPD